CLINICAL TRIAL: NCT02711852
Title: A Long-term, Continued Treatment and Follow-up Study in Subjects With Hematologic Malignancies Treated With Duvelisib (IPI-145)
Brief Title: A Long-term, Continued Treatment and Follow-up Study in Participants With Hematologic Malignancies Treated With Duvelisib (IPI-145)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-23
Record Dates: First submitted 2016-03-15; First posted 2016-03-17 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Duvelisib (Experimental): Participants received the same dose from their previous duvelisib study. All doses were taken twice daily. Two dose reductions were allowed per participant, but doses were not less than 10 milligrams (mg). Participants received duvelisib until disease progression or unacceptable toxicity.
  Interventions: Drug: Duvelisib

INTERVENTIONS:
Drug: Duvelisib — Administered as oral capsules
  Other Names: IPI-145; VS-0145; COPIKTRA

SUMMARY:
This was a long-term, continued treatment study that evaluated the long-term safety, clinical activity, and overall survival (OS) of duvelisib in individuals with hematologic malignancies that were previously treated with duvelisib in a previous sponsor-approved study.

DETAILED DESCRIPTION:
Study IPI-145-23 was an international, multicenter, open-label, single-arm, Phase 2 study designed to evaluate the long-term safety, clinical activity, and overall survival data of duvelisib in individuals with hematologic malignancies. Only individuals who have participated in a previous duvelisib study that were approved by the sponsor were allowed to enroll in the study.

Participants in active treatment and participants in survival follow-up were allowed to rollover to this study. For participants on active treatment, participants continued the same dose from their previous duvelisib study administered twice daily for 28-day continuous cycles until disease progression or unacceptable toxicity and then followed in a survival follow-up period. For participants in survival follow-up, participants continued to be followed-up for survival in this study for the duration as outlined in their previous duvelisib study.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in a previous study of duvelisib, and:

  * Be actively receiving duvelisib monotherapy on the previous study (within 14 days of study entry) and demonstrating clinical benefit (complete response [CR]/ partial response [PR]/ stable disease [SD]) of continued use, or
  * Be in the survival follow-up phase of a previous duvelisib study
* Have completed the required components of the previous study and be appropriate for enrollment into this long-term continued treatment and follow-up study, as determined by the Sponsor

Exclusion Criteria:

* Had any ongoing ≥ Grade 3 adverse event (AE) considered related to duvelisib treatment at screening
* Was pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Denver, Colorado
  - Sarasota, Florida
  - Nashville, Tennessee
  - UT MD Anderson Cancer Center, Houston, Texas
- Azienda Ospedaliera Santa Maria di Terni/SC Oncoematologia, Terni, Umbria, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 19 participants were enrolled in the current study from 3 previous studies: IPI-145-01(NCT01549106), IPI-145-02 (NCT01476657), and IPI-145-08 (NCT02204982).
Groups:
- Duvelisib: Oral capsules administered twice daily. Participants continued to receive the same dose level as their previous duvelisib study.
Period: Overall Study
Arm/Group | Duvelisib
Started | 19
Received At Least 1 Dose of Study Drug | 19
Completed | 9
Not Completed | 10
Not completed — Death | 5
Not completed — Lost to Follow-up | 1
Not completed — Completed follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All Treated Analysis Set included all participants who received at least one dose of duvelisib.
Arm/Group | Duvelisib
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to 45 months
Population: All Treated Analysis Set included all participants who received at least one dose of duvelisib.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib
Number analyzed (Participants) | 19
Participants | 17

2. Secondary Outcome: Best Overall Response (BOR) to Duvelisib as Assessed by the Investigator
Description: There were no formal secondary endpoints planned and captured data was based on disease response assessment and overall survival (OS) as defined in the participant's previous study.
  BOR was defined as the best time point response that a participant achieves during the study, with the response ranked according to the following order (from best to worst): complete response (CR), complete response with incomplete marrow recovery (CRi), partial response (PR), stable disease (SD).
Time Frame: Up to 45 months
Population: All Treated Analysis Set included all participants who received at least one dose of duvelisib and for whom a documented response was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib
Number analyzed (Participants) | 16
Participants
  CR/CRi | 9
  PR | 5
  SD | 1
  Response not evaluable | 1

3. Secondary Outcome: Overall Survival (OS)
Description: No formal secondary endpoints were planned for this study. OS was monitored in participants who continued to receive duvelisib treatment and/or in the long-term survival follow-up period in a previous duvelisib study and the number of participants alive at end of study were reported.
  Participants being followed for OS were contacted by the study site approximately every 6 months to collect survival status and data pertaining to any other alternative antineoplastic therapy.
Time Frame: Up to 45 months
Population: All Treated Analysis Set included all participants who received at least one dose of duvelisib.
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib
Number analyzed (Participants) | 19
Participants | 14

ADVERSE EVENTS:
Time Frame: Up to 45 months
Description: All Treated Analysis Set included all participants who received at least one dose of duvelisib. All-cause mortality, serious adverse event, and other adverse event data were pre-specified to be collected as a single arm for any participant who received at least one dose of the study drug, regardless of their dose level.
Arm/Group | Duvelisib
All-Cause Mortality (participants affected / at risk) | 5/19
Serious Adverse Events (participants affected / at risk) | 5/19
Other Adverse Events (participants affected / at risk) | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=19)
Diarrhoea (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=19)
Anaemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Reflux gastritis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 4
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Brucellosis (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Blood triglycerides increased (Investigations) | 1
Lipase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Weight decreased (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Skin fragility (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02711852/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT02711852/SAP_001.pdf